CLINICAL TRIAL: NCT00644176
Title: A Randomized, Open Label, Clinical Trial of the Pharmacokinetics of Azithromycin in Serum, Bronchial Washings and Lung Tissue Following a Single Dose of Azithromycin Sustained Release (2 Gram) or Commercial Azithromycin Tablet (500 mg) to Cancer Patients That Require Lung Resection
Brief Title: A Randomized, Open Label, Clinical Trial of the Pharmacokinetics of Azithromycin Following a Single Dose of Azithromycin Sustained Release (2 Gram) or Commercial Azithromycin Tablet (500 mg) to Cancer Patients That Require Lung Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A0661145
Record Dates: First submitted 2008-03-19; First posted 2008-03-26 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: azithromycin immediate release (Zithromax); Other: placebo
- 2 (Experimental)
  Interventions: Drug: azithromycin SR; Other: placebo

INTERVENTIONS:
Drug: azithromycin immediate release (Zithromax) — azithromycin IR 500 mg tablet by mouth for 1 dose
  Arms: 1
Other: placebo — placebo
  Arms: 1
Drug: azithromycin SR — 2.0 g by mouth in the form of liquid for 1 dose
  Arms: 2
Other: placebo — placebo
  Arms: 2

SUMMARY:
The objective of this trial was to characterize the pharmacokinetics of the currently marketed azithromycin immediate release tablet formulation (AZ-IR) versus the azithromycin sustained release liquid formulation (AZ-SR) in lung tissue and bronchial washings, the latter consisting of the epithelial lining fluid (ELF) and cellular elements, mainly alveolar macrophages (AM).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were hospitalized subjects diagnosed with lung cancer that had consented to surgery requiring lung resection who had a life expectancy of >6 months.

Exclusion Criteria:

Key exclusion criteria were antibiotic prophylaxis prior to surgery, diffuse, non-infectious lung disease, history of cigarette smoking of >5 packs per year, patients with any infectious disease that required antibiotic therapy, administration of drugs known to interfere with azithromycin pharmacokinetics, and subjects on chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2004-11; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Azithromycin Cmax, Tmax, AUC72, (or AUClast for serum) and AUC24 from serum | predose, and at and at 2, 4, 8, 12, 16, 24, 48, and 72 hours postdose
Azithromycin Cmax, Tmax, AUC72, and AUC24 in epithelial lining fluid and alveolar cells from bronchoalveolar lavage and lung tissue samples | 2, 4, 8, 12, 16, 24, 48, and 72 hours postdose

SECONDARY OUTCOMES:
12-lead electrocardiograms (ECGs) | Screening and 72 hours postdose
adverse events (AEs) | Treatment day 0, and at 2, 4, 8, 12, 16, 24, 48, and 72 hours postdose
safety laboratory tests | Treatment day 0 and 72 hours postdose
vital signs | Screening and Treatment day 0

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Pisa, Italy

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661145&StudyName=A%20Randomized%2C%20Open%20Label%2C%20Clinical%20Trial%20of%20the%20Pharmacokinetics%20of%20Azithromycin%20Following%20a%20Single%20Dose%20of%20Azithromycin%20Sustained%20Rel